CLINICAL TRIAL: NCT02118961
Title: Confirmatory Study to Evaluate the Immunogenicity of Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed (DTaP Vaccine, BK1301) as a Booster in Adolescents
Brief Title: Study of BK1301 (DTaP Vaccine) as a Booster in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: The Research Foundation for Microbial Diseases of Osaka University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BKD1A
Record Dates: First submitted 2014-04-13; First posted 2014-04-21 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: Diphtheria; Tetanus; Pertussis; DTaP vaccine; Adolescents
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Tetanus Toxoid; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BK1301 (Experimental)
  Interventions: Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed (DTaP vaccine, BK1301)
- DT toxoid (Active Comparator)
  Interventions: Biological: Adsorbed Diphtheria-Tetanus Combined Toxoid (DT toxoid)

INTERVENTIONS:
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed (DTaP vaccine, BK1301) — 0.5 mL, subcutaneous injection
  Other Names: TRIBIK®
  Arms: BK1301
Biological: Adsorbed Diphtheria-Tetanus Combined Toxoid (DT toxoid) — 0.1 mL, subcutaneous injection
  Other Names: DTBIK®
  Arms: DT toxoid

SUMMARY:
This study is designed to assess the immunogenicity and safety of DTaP vaccine (BK1301) as a booster dose in adolescents.

The purposes of this study are as follows:

* To confirm the non-inferiority of BK1301 to Adsorbed Diphtheria-Tetanus Combined Toxoid (DT toxoid) with respect to booster responses for anti-diphtheria toxoid (anti-D) and anti-tetanus toxoid (anti-T) antibodies
* To confirm that booster responses for anti-pertussis toxoid (anti-PT) and anti-Filamentous Hemagglutinin (anti-FHA) antibodies are more than 80% of participants received BK1301

ELIGIBILITY:
Inclusion Criteria:

* Age 11 or 12 years on the day of injection
* Received 3 or 4 doses of DTaP vaccine

Exclusion Criteria:

* History of pertussis, diphtheria, tetanus
* History of anaphylaxis to vaccine components
* Serious conditions or diseases of the heart, vein, blood, respiratory, hepar, kidney, digestive system, psychiatric or nervous system
* Transfused or received gamma globulin within 3 months, or received high-dose gamma globulin within 6 months before the day of injection

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 446 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shintaro Okada, M.D., Ph.D., Study Director — Osaka University
Locations (7):
- Japan (7):
  - Investigational site, Fukuoka, Fukuoka
  - Investigational site, Itoshima-shi, Fukuoka
  - Investigational site, Kasuga-shi, Fukuoka
  - Investigational site, Hiroshima, Hiroshima
  - Inverstigational site, Kumagaya-shi, Saitama
  - Investigational site, Shizuoka, Shizuoka
  - Inverstigational site, Shinjuku-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BK1301 | DT Toxoid
Started | 224 | 222
Completed | 223 | 222
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BK1301 | DT Toxoid | Total
Number analyzed (Participants) | 224 | 222 | 446
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 224 | 222 | 446
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 104 | 217
  Male | 111 | 118 | 229

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Booster Responses for Anti-diphtheria Toxoid (Anti-D) and Anti-tetanus Toxoid (Anti-T) Antibodies
Description: Booster response was defined as post titer ≥ 0.4 IU/mL and post/pre titer ≥ 4 increase.
Time Frame: pre-vaccination and 28-42 days after vaccination
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | BK1301 | DT Toxoid
Number analyzed (Participants) | 223 | 222
percentage of Participants
  anti-D | 100.0 [98.4 to 100.0] | 99.5 [97.5 to 100.0]
  anti-T | 98.7 [96.1 to 99.7] | 97.3 [94.2 to 99.0]

2. Primary Outcome: Percentage of Participants With Booster Responses for Anti-pertussis Toxoid (Anti-PT) and Anti-Filamentous Hemagglutinin (Anti-FHA) Antibodies
Description: Booster response was defined as post titer ≥ 20 EU/mL and post/pre titer ≥ 4 increase in a subject with pre titer < 20 EU/mL, or post/pre titer ≥ 2 increase in a subject with pre titer ≥ 20 EU/mL.
Time Frame: pre-vaccination and 28-42 days after vaccination
Population: The Outcome Measure was only pre-specified for the BK1301 Arm/Group.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | BK1301
Number analyzed (Participants) | 223
percentage of Participants
  anti-PT | 91.0 [86.5 to 94.4]
  anti-FHA | 91.5 [87.0 to 94.8]

3. Secondary Outcome: Percentage of Participants With Anti-D and Anti-T Antibody Titers Above Protocol Defined Cut-off Values
Description: Protocol defined cut-off values were 0.1 IU/mL for anti-D and 0.01 IU/mL for anti-T.
Time Frame: 28-42 days after vaccination
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | BK1301 | DT Toxoid
Number analyzed (Participants) | 223 | 222
percentage of Participants
  anti-D | 100.0 [98.4 to 100.0] | 100.0 [98.4 to 100.0]
  anti-T | 100.0 [98.4 to 100.0] | 100.0 [98.4 to 100.0]

4. Secondary Outcome: Percentage of Participants With Anti-PT and Anti-FHA Antibody Titers Above Protocol Defined Cut-off Values
Description: Protocol defined cut-off values were 10 EU/mL.
Time Frame: 28-42 days after vaccination
Population: The Outcome Measure was only pre-specified for the BK1301 Arm/Group.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | BK1301
Number analyzed (Participants) | 223
percentage of Participants
  anti-PT | 100.0 [98.4 to 100.0]
  anti-FHA | 100.0 [98.4 to 100.0]

5. Secondary Outcome: Geometric Mean Titers (GMTs) of Anti-D and Anti-T Antibodies
Time Frame: 28-42 days after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1301 | DT Toxoid
Number analyzed (Participants) | 223 | 222
IU/mL
  anti-D | 20.856 [18.221 to 23.872] | 15.581 [13.748 to 17.658]
  anti-T | 13.378 [11.838 to 15.118] | 11.638 [10.348 to 13.090]

6. Secondary Outcome: Geometric Mean Titers (GMTs) of Anti-PT and Anti-FHA Antibodies
Time Frame: 28-42 days after vaccination
Population: The Outcome Measure was only pre-specified for the BK1301 Arm/Group.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1301
Number analyzed (Participants) | 223
EU/mL
  anti-PT | 241.15 [210.65 to 276.07]
  anti-FHA | 344.46 [309.72 to 383.10]

7. Secondary Outcome: Geometric Mean Titer Ratios of Anti-D and Anti-T Antibodies
Description: Ratios were calculated as 28-42 days after vaccination titers over pre vaccination titers
Time Frame: pre vaccination and 28-42 days after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: titer ratio
Arm/Group | BK1301 | DT Toxoid
Number analyzed (Participants) | 223 | 222
titer ratio
  anti-D | 137.5 [107.8 to 175.5] | 106.3 [83.9 to 134.7]
  anti-T | 47.9 [38.9 to 59.0] | 44.3 [36.4 to 53.9]

8. Secondary Outcome: Geometric Mean Titer Ratios of Anti-PT and Anti-FHA Antibodies
Description: Ratios were calculated as 28-42 days after vaccination titers over pre vaccination titers
Time Frame: pre vaccination and 28-42 days after vaccination
Population: The Outcome Measure was only pre-specified for the BK1301 Arm/Group.
Measure: Geometric Mean (95% Confidence Interval); unit: titer ratio
Arm/Group | BK1301
Number analyzed (Participants) | 223
titer ratio
  anti-PT | 12.6 [10.5 to 15.2]
  anti-FHA | 8.5 [7.2 to 10.0]

9. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: 28-42 days following vaccination
Measure: Number; unit: percentage of participants
Arm/Group | BK1301 | DT Toxoid
Number analyzed (Participants) | 223 | 222
percentage of participants | 90.1 | 89.6

ADVERSE EVENTS:
Arm/Group | BK1301 | DT Toxoid
Serious Adverse Events (participants affected / at risk) | 0/223 | 0/222
Other Adverse Events (participants affected / at risk) | 200/223 | 194/222
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BK1301 (N=223) | DT Toxoid (N=222)
Injection site erythema (General disorders) | 167 | 160
Injection site induration (General disorders) | 95 | 84
Injection site pain (General disorders) | 125 | 85
Injection site pruritus (General disorders) | 132 | 113
Injection site swelling (General disorders) | 162 | 148
Injection site warmth (General disorders) | 115 | 87
Pyrexia (General disorders) | 15 | 3
Nasopharyngitis (Infections and infestations) | 12 | 15
Headache (Nervous system disorders) | 17 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other